CLINICAL TRIAL: NCT04397627
Title: Enhanced Recovery Pathways, Patient-reported Outcomes and Return to Intended Oncological Therapy After Colorectal Surgery: the Italian ColoRectal Anastomotic Leakage Study Group (iCral 3).
Brief Title: ERAS Program Items Adherence, PROMs and RIOT After Colorectal Surgery
Acronym: iCral3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ospedale C & G Mazzoni (Other)
Responsible Party: Principal Investigator, Marco Catarci, MD, FACS; Director, General Surgery Unit, Ospedale C & G Mazzoni
Other Study IDs: iCral3
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Surgery; Enhanced Recovery After Surgery; Patient Reported Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colorectal resection — All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after written informed consent.

SUMMARY:
Prospective multicenter observational no-profit study evaluating the impact of ERAS program items adherence rates on patient-reported outcomes (PRO) and return to intendend oncologic therapy (RIOT) after colorectal resection.

Prospective enrollment from November 2020 to October 2021 in 60 Italian surgical centers. All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after written informed consent. A total of 3,000 patients is expected based on a mean of 50 cases per center.

DETAILED DESCRIPTION:
BACKGROUND Enhanced Recovery After Surgery (ERAS) is a multimodal and multifactorial approach to the optimization of perioperative management. In order to modify and improve the response to surgery-induced trauma, the program relies on a series of evidence-based items related to pre-, intra- and post-operative care. Several meta-analyses on ERAS showed a significant reduction of morbidity rates and length of stay after colorectal surgery. However, program implementation outside clinical trials is still extremely variable, as the necessary multidisciplinary involvement makes the program vulnerable to various areas of failure, that explain the great variation in adherence rates to program items.

During the early phase of program implementation, adherence rate to program items rarely goes beyond 50%, needing to reach at least 70% in order to significantly improve results (faster recovery and reduced morbidity). Recent cohort studies reported a mean adherence rate to ERAS items between 63 and 75%. In other studies, adherence to ERAS items was higher, reaching up to 90%. Moreover, a clear and significant dose-effect curve between adherence rate to ERAS program items and early outcomes was demonstrated, and recent evidence deriving from retrospective studies suggests that ERAS programs may also offer a definite advantage over long-term survival after colorectal resection for malignancy. While many studies to date have focused on early outcomes (i.e. earlier return of bowel function, lower complication rates, and/or shorter length of inpatient stay), for the majority of oncologic operations, however, postoperative recovery carries the additional demand of returning the patient to adjuvant oncologic therapies. It is still unclear if ERAS program could improve the failure to "return to intended oncologic therapy" (RIOT) after cancer surgery due to complications and lingering poor performance status, that is strongly associated with worse oncologic outcomes, including shortened overall survival. Measuring patient-reported outcomes (PROs) addresses the gap in enhanced recovery assessment by incorporation of patient-centered quality into our global assessment of outcomes. Taken together, these data establish a paradigm for association of perioperative medical care to long-term oncologic outcomes-revealing how the perioperative care team's actions over a relatively short number of days and hours around the time of a cancer surgery can improve cancer-specific survival. The concept is that various perioperative techniques, protocols, and agents will blunt the patient's perioperative stress response, reduce complications, and improve functional recovery after surgery. Together, these effects allow more people to RIOT in a more timely fashion and in a more complete way. To the extent that the combination of preservation of immune competence and more reliable return to adjuvant therapies then reduce recurrence rates, longer and more meaningful survivals may be achieved.

Therefore, the Italian Colorectal Anastomotic Leakage study group planned this study to prospectively evaluate the impact of adherence to ERAS program items after colorectal resections on PRO in the whole population and on failure to RIOT for malignant disease.

Outcome measures

1. Preoperative risk factors (age, gender, obesity, nutritional status, diabetes, cardiovascular disease, chronic liver disease, renal failure, inflammatory bowel disease, perioperative steroid therapy, ASA class I-II vs III, SARS-CoV-2 infection)
2. Operative parameters (approach, procedure, anastomotic technique, length of operation, pTNM stage)
3. Adherence to ERAS program items

Primary Endpoints

1. Patient-related outcomes measures (PROMs):
2. Return to intended oncologic therapy (RIOT)

   Secondary Endpoints
3. Anastomotic leakage rate
4. Minor and major complication rates
5. Overall length of postoperative hospital stay (including any readmission)
6. Readmission and reoperation rates

Recorded data and follow-up During the postoperative period, the local attending surgeon will make any decision for complementary exams and imaging according to his own criteria, the only exception being the creation of a proximal diverting stoma at operation, that mandates routine check of anastomotic integrity through an intraluminal contrast exam (standard x-rays or CT scan) three to six weeks after the operation. The rate of any complication will be calculated and graded according to Clavien-Dindo including all anastomotic leaks, wound infection (according to the definitions of the Centers for Disease Control and Prevention and wound culture), pneumonia (clinical symptoms, and physical and radiological examinations), central line infection (positive blood culture), urinary tract infection (positive urine culture with bacterial count). Patients will be followed-up in the outpatient clinic up to 8 weeks after discharge from the hospital.

Anastomotic dehiscence (any deviation from the planned postoperative course related to the anastomosis, or presence of pus or enteric contents within the drains, presence of abdominal or pelvic collection in the area of the anastomosis on postoperative CT scan, leakage of contrast through the anastomosis during enema or evident anastomotic dehiscence at reoperation for postoperative peritonitis) will be defined and graded according to international consensus guidelines. Anastomotic testing will be performed intraoperatively with the air-leak test (ALT) and using ICG-NIR-NBI with a standard protocol [ICG 25 mg diluted in 10 mL saline (2.5 mg/mL); first bolus i.v. injection of 4 mL (10 mg) after vascular control and mesenteric division, just before proximal and/or distal bowel division; second bolus i.v. injection of 4 mL (10 mg) just before joining anastomotic stumps; third (optional) bolus i.v. injection of 2 mL (5 mg) after the anastomosis is completed; NIR-NBI observation within 60-120" after every ICG injection (direct, laparoscopic or endoscopic)].

PROM questionnaires will be administered to all enrolled patients four to one week before the planned operation, on the day of discharge (or POD5), and 6 weeks after the operation.

RIOT rates will be recorded in all patients submitted to surgery for malignancy, according to national guidelines for colorectal cancer.

After anonymization, all data of each single case will be prospectively uploaded by local investigator(s) on a protected web-based database and incorporated into a spreadsheet for data analysis, checking for any discrepancy, that will be addressed and solved through strict cooperation between chief investigator, data manager and participating centers.

This study protocol will be submitted to the coordinating center ethics committee (Comitato Etico Regionale delle Marche - C.E.R.M.) for approval and then registered at ClinicalTrials.gov. Thereafter, all the participating centers will obtain authorization to participate from the local institutional review board. Anonymized participant-level datasets will be available after study completion upon reasonable request by contacting the principal investigator.

Statistical Analysis Quantitative values will be expressed as mean ± standard deviation (SD), median and range; categorical data with percentage frequencies. For categorical data, analysis will include the use of cross tabulation, chi squared or Fisher's exact test where indicated. Continues or discrete variables will be analyzed using Student's two-sided t test (allowing for heterogeneity of variances) or with a non-parametric test (Mann-Whitney U test or Kruskal-Wallis test as indicated). Joint and conditional multivariate association between all variables shown to be significant on univariate analysis will be assessed using binary logistic or multiple linear regression. The odds ratio (OR) will be presented followed by 95% confidence interval (95% CI). Concerning comparison of nutritional status scores, areas under the receiver-operating characteristics curve (AUC-ROC) will be calculated for all endpoints, considering values from 0.7 to 0.8 as acceptable, 0.8 to 0.9 excellent, and above 0.9 as outstanding (40). Differences in AUC-ROC curves will be analyzed with the chi-squared test. Optimal cut-off points will be obtained applying Youden's Index (Sensitivity+Specificity-1), choosing those values of the AUC-ROC curve where this index is maximal. Negative predictive values (NPV) and positive predictive values (PPV) will also be calculated; finally, a logistic regression model will be built using the presence/absence of endpoint as dependent variable, and nutritional scores ≤ or > the cut-off values as explanatory factors; using logistic transformation of the linear predictors, the probabilities of the endpoint related to the different combinations of factors level will be obtained . For all statistical tests the significant level is fixed at p < .05. Statistical analyses will be carried out using STATA software (Stata Corp. College Station, Texas, USA).

Sample size Adherence to at least 70% of the ERAS program items was identified as a cut-off for significant improvement of outcomes , with a 2:1 expected ratio below:above the cut-off. Estimating a reduction of postoperative PRO from preoperative baseline (1.0) at 0.7 for adherence above the cut-off and at 0.64 for adherence below the cut-off, alpha 0.04, beta 0.8, the required sample size is n=2,406 (802 cases above 70% adherence and 1,604 below 70% adherence). Reported rates for failure to RIOT and ERAS program items adherence below or above 70% are 13 and 6.5%, respectively (27); the required sample size for evaluation of failure to RIOT is n=885 (295 cases above 70% adherence and 590 below 70% adherence). Based on previous iCral observational study on colorectal surgery in Italy, the expected ratio of malignant:benign indications to surgery is 70:30 (2,100 resections for malignancy and 900 resections for benign disease on the basis of 3,000 expected cases).

ELIGIBILITY:
Inclusion Criteria:

1. Patients submitted to laparoscopic/robotic/open/converted ileo-colo-rectal resection with anastomosis, including planned Hartmann's reversals.
2. American Society of Anesthesiologists' (ASA) class I, II or III
3. Elective or delayed urgency surgery
4. Patients' written acceptance to be included in the study.

Exclusion Criteria:

1. American Society of Anesthesiologists' (ASA) class IV-V
2. Emergent surgery
3. Pregnancy
4. Hyperthermic intraperitoneal chemotherapy for carcinomatosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing elective colorectal surgery with anastomosis will be included in a prospective database after written informed consent.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported outcome measure #1; Health Questionnaire; Euro-QoL Group EQ-5D-5L™; | Before the operation, postoperative day 5, 4 to 6 weeks after the operation
  Quality of life questionnaire based on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Scores ranging from 5 (worst) to 125 (best)
Change in patient-reported outcome measure #2; Health Questionnaire: MD Anderson Symptom Inventory for gastrointestinal surgery patients (MDASI-GI) | Before the operation, postoperative day 5, 4 to 6 weeks after the operation
  Specific quality of life questionnaire for patients submitted to GI surgery: based on 24 questions with scores ranging from 0 (best) to 10 (worst); total score from 0 (best) to 240 (worst)
Change in patient-reported outcome measure #3; Health Questionnaire Functional Assessment of Cancer Therapy - Colorectal® (FACT-C) | Before the operation, postoperative day 5, 4 to 6 weeks after the operation
  Specific quality of life questionnaire for patients with colorectal cancer. Scores ranging form 0 (worst) to 144 (best).
Return to intended oncologic therapy (RIOT) | 8 weeks after the operation
  Number of patients eligible for adjuvant therapy after surgery for colorectal cancer that receive appropriate treatment starting within 8 weeks after the operation

SECONDARY OUTCOMES:
Anastomotic leakage rate | within 8 weeks from operation
  number of anastomotic leakage
Overall morbidity rate | within 8 weeks from operation
  number of any perioperative adverse event graded according to Clavien-Dindo
Major morbidity rate | within 8 weeks from operation
  number of Clavien-Dindo grade >II perioperative adverse events
Length of hospital stay (LOS) | within 8 weeks from operation
  Total number of days spent in the hospital (including any readmission)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Catarci, MD, FACS, Principal Investigator — Ospedale CG Mazzoni Ascoli Piceno
Locations (8):
- Italy (8):
  - UOC Chirurgia Generale Universitaria - Ospedale San Salvatore - L'Aquila, L’Aquila, AQ
  - S.C. Chirurgia Generale e Oncologica - Azienda Ospedaliera S. Croce e Carle - Cuneo, Italia, Cuneo, CN
  - UOC Chirurgia Generale ad Indirizzo Oncologico - IRCCS San Martino IST - Genova, Genova, GE
  - UOC Chirurgia Generale - Ospedale di Esine (BS) - ASST Valcamonica, Esine, NS
  - UOC Chirurgia Generale e D'Urgenza . Azienda Ospedaliera San Camillo Forlanini Roma, Roma, RM
  - UOC Chirurgia Generale - Ospedale Sacro Cuore Don Calabria Negrar Verona, Negrar, VR
  - U.O.C. di Chirurgia Generale e dell'Esofago e Stomaco - AOUI di Verona, Verona, VR
  - SOC Chirurgia Colorettale - Istituto Nazionale dei Tumori - IRCCS Fondazione "G.Pascale" - Napoli, Napoli

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Background] Kehlet H. Fast-track colorectal surgery. Lancet. 2008 Mar 8;371(9615):791-3. doi: 10.1016/S0140-6736(08)60357-8. No abstract available. PMID 18328911
- [Background] Aloia TA, Zimmitti G, Conrad C, Gottumukalla V, Kopetz S, Vauthey JN. Return to intended oncologic treatment (RIOT): a novel metric for evaluating the quality of oncosurgical therapy for malignancy. J Surg Oncol. 2014 Aug;110(2):107-14. doi: 10.1002/jso.23626. Epub 2014 May 21. PMID 24846705
- [Background] Italian ColoRectal Anastomotic Leakage (iCral) Study Group. Anastomotic leakage after elective colorectal surgery: a prospective multicentre observational study on use of the Dutch leakage score, serum procalcitonin and serum C-reactive protein for diagnosis. BJS Open. 2020 Jun;4(3):499-507. doi: 10.1002/bjs5.50269. Epub 2020 Mar 5. PMID 32134216